CLINICAL TRIAL: NCT06715501
Title: Efficacy and Safety of Cadonilimab Combined with Chemoradiotherapy in Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma-A Single-arm Exploratory Study
Brief Title: Efficacy and Safety of Cadonilimab and Chemoradiotherapy in Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Taoqingsong, chief physician, Ningbo No. 1 Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-E-0195
Record Dates: First submitted 2024-11-21; First posted 2024-12-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma; II-IIIB Stages
Keywords: locally advanced ESCC; II-IIIB stage; Cadonilimab; Chemoradiotherapy
MeSH Terms: interventions — Radiotherapy; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cadonilimab combined with Chemoradiotherapy (Experimental): Patients with advanced unresectable esophageal squamous cell carcinoma who meet the criteria, will first receive induction therapy with cetuximab combined with paclitaxel and carboplatin chemotherapy for 2 cycles. Within 3 weeks after the second dose, RECIST v1.1 will be used for clinical tumor imaging evaluation. Patients without progression will further receive synchronous radiotherapy and chemotherapy.
  PTV-C accepts 50.4Gy, 28 times; Radiotherapy combined with paclitaxel and carboplatin weekly regimen. Within three months after completion, conduct safety assessments and preliminary evaluations of tumor response every three weeks. Consolidate treatment with cetuximab until 1 year or intolerance or disease progression occurs.
  Interventions: Drug: Cadonilimab; Radiation: radiotherapy; Drug: carboplatin, paclitaxel

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab is a PD-1/CTLA-4 bispecific antibody. The drug is administered at a fixed dose of 10mg/kg, intravenously (i.v.), on day 1, every 3 weeks (q3w), until disease progression or intolerable toxicity occurs, with a maximum treatment duration of 1 year.
Radiation: radiotherapy — GTV is defined as visible lesions (GTVp: primary lesion; GTVn: metastatic lymph nodes), CTVp is defined as 3cm above and below the primary lesion, with 0.5cm outward expansion around the periphery, and CTVn is defined as 0.5cm outward expansion of GTVn; PTVp is an outward expansion of 0.5cm for CTVp, and PTVn is an outward expansion of 0.5cm for CTVn. Radiotherapy dose: DT50.4Gy/28f, once daily, 5 times a week
Drug: carboplatin, paclitaxel — Induction chemotherapy: carboplatin 5AUC，q3w; Paclitaxel 135mg/m2,q3w. Simultaneous chemotherapy: 2AUC/W，total 5w; Paclitaxel 50mg/m2/w，total 5w

SUMMARY:
This study is a single center, prospective, single arm exploratory clinical trial aimed at evaluating the efficacy and safety of sequential chemoradiotherapy combined with cetuximab in unresectable locally advanced esophageal squamous cell carcinoma.

Patients with advanced unresectable esophageal squamous cell carcinoma who meet the criteria, after signing the informed consent form, will first receive induction therapy with cetuximab combined with paclitaxel and carboplatin chemotherapy for 2 cycles. Within 3 weeks after the second dose, RECIST v1.1 will be used for clinical tumor imaging evaluation, and if necessary, gastroscopy biopsy will be performed. Patients without progression will further receive synchronous radiotherapy and chemotherapy.

PTV-C accepts 50.4Gy, 28 times; Radiotherapy combined with paclitaxel and carboplatin weekly regimen. Within three months after completion, conduct safety assessments and preliminary evaluations of tumor response every three weeks. Consolidate treatment with cetuximab until 1 year or intolerance or disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of locally advanced esophageal squamous cell carcinoma (TN+M0 or T2-3NxM0) by histological examination and/or cytological examination；
* TNM clinical stage II-IIIB that cannot be surgically resected ;
* ECOG score 0-1 points;
* Expected survival ≥ 6 months;
* Without anti-tumor treatment in the past (including but not limited to surgery, radiotherapy, chemotherapy, anti vascular therapy, immunotherapy, etc.);
* Pathological specimens available;
* At least one measurable target lesion or pathological enlargement of lymph nodes with a single lymph node CT scan short diameter ≥ 15mm (according to the efficacy evaluation criteria for solid tumors RECIST 1.1) ;
* The main organ functions well and meets the following standards:

  1. Blood routine examination (without blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days): hemoglobin (Hb) ≥ 90 g/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 80 × 109/L;
  2. Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Serum total bilirubin (TBIL) ≤ 1.5 × ULN (Gilbert syndrome subjects, ≤ 3 × ULN); Serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance rate ≥ 60mL/min;
  3. Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
* Subjects with fertility must use appropriate contraception methods during the study period and within 120 days after the last dose. They must have a negative serum pregnancy test within 7 days before enrollment and must be non lactating subjects.

Exclusion Criteria:

* Other malignant tumors within 5 years prior to the start of this study;
* High risk of gastrointestinal bleeding, esophageal fistula or perforation;
* Unrelieved toxic reactions of grade ≥ 1(excluding alopecia and fatigue; hematological toxicity must be recovered to grade ≤1 or baseline before enrollment);
* Weight loss of ≥20% within 90 days prior to signing the informed consent form;
* Poor nutritional status or a PG-SGA score of ≥9;
* Any severe and/or uncontrolled diseases. This includes:

  1. Uncontrolled blood pressure (systolic pressure ≥150mmHg or diastolic pressure ≥100mmHg);
  2. Suffering from grade ≥2 myocardial ischemia or myocardial infarction, arrhythmia (QTc ≥470ms), and grade ≥2 congestive heart failure (New York Heart Association [NYHA] classification);
  3. History of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, or other uncontrolled acute pulmonary diseases;
  4. Active or uncontrolled severe infections (grade ≥2 CTCAE infections);
  5. Liver cirrhosis, active hepatitis; active hepatitis (for hepatitis B: positive HBsAg and HBV DNA levels exceeding the upper limit of normal; for hepatitis C: positive HCV antibodies and HCV viral load exceeding the upper limit of normal);
  6. Active syphilis;
  7. Renal failure requiring hemodialysis or peritoneal dialysis;
  8. A history of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* Poorly controlled diabetes (fasting blood glucose [FBG] > 10mmol/L);
* Major surgical treatment, incisional biopsy, or significant traumatic injury within 60 days before the start of the study; or long-term unhealed wounds or fractures;
* Serious arterial/venous thrombotic events within 6 months before the start of the study, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
* A history of substance abuse and inability to quit or with mental disorders;
* Tumor-related symptoms and treatments:

  1. Thoracic radiotherapy;
  2. Traditional Chinese medicine drugs approved by the NMPA with clear anti-tumor indications in the drug instructions within 2 weeks before the start of the study (including Compound Esophageal Cancer Capsules, Kangai Injection, Kanglaite Capsules/Injection, Aidi Injection, Bitternut Oil Injection/Capsules, Xiaoai Ping Tablets/Injection, Huachansu Capsules, etc.);
  3. Uncontrollable, repeatedly drained pleural effusion, pericardial effusion, or ascites (investigator's judgment);
  4. Central nervous system metastasis and/or meningeal carcinomatosis;
* Study treatment-related:

  1. History of attenuated live vaccine administration within 14 days before the start of the study or plans for attenuated live vaccine administration during the study;
  2. Severe hypersensitivity reactions after the use of monoclonal antibodies;
  3. Active autoimmune diseases requiring systemic treatment (such as disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years before the start of the study, excluding replacement therapies (e.g., thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency);
  4. Immunodeficiency or receiving systemic glucocorticoid treatment or any other form of immunosuppressive therapy (dose >10mg/day prednisone or other equivalent hormones) and still in use within 2 weeks of the first administration;
  5. A history of active tuberculosis;
* Participation in other clinical studies within 4 weeks before the start of the study;
* A history of severe allergies;
* Allergic to the active ingredients or excipients of the study drugs, such as camrelizumab, paclitaxel, carboplatin, etc.;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival rate | 2 year after the end of treatment
Incidence of Treatment-Emergent Adverse Events | Within three months after radiotherapy
  The incidence of adverse events (AE) and serious adverse events (SAE) within three months after radiotherapy, and the incidence of treatment termination caused by AE/SAE

SECONDARY OUTCOMES:
Progression free survival (PFS) | From the randomization date until the first recorded date of progression or death from any cause, whichever comes first, assessed up to 36 months
Overall survival (OS) | From the randomization date until death from any cause，assessed up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided